# USE OF NORETHINDRONE ACETATE FOR MANAGEMENT OF BLEEDING ASSOCIATED WITH THE ETONOGESTREL CONTRACEPTIVE IMPLANT

Katherine McCracken, Scott LaJoie, Meredith Loveless, S. Paige Hertweck, Rachael Polis, Margaret Abraham

Norton Children's Gynecology, University of Louisville, Louisville, KY

#### **HYPOTHESIS:**

Oral progesterone is a useful therapy for the management of bleeding associated with the etonogestrel contraceptive implant.

### **OBJECTIVE:**

The overall objective of this study is to confirm that oral progesterone is an effective way to manage bothersome bleeding; thus increasing the rate of continuation of the etonogestrel contraceptive implant in adolescents.

#### **BACKGROUND AND SIGNIFICANCE:**

Of the approximately three million pregnancies annually in the United States, 50 percent are unintended pregnancies. Adolescents bear a significant burden of such unintended pregnancies, with 82 percent of adolescent pregnancies being unplanned (1). It is well documented that adolescent pregnancies have deleterious effects on women's health and educational attainment, the health of newborns, and incur a significant emotional and financial burden, both for the individual and society as a whole. Furthermore, greater than one-third of unintended adolescent pregnancies end in abortion (2).

While most sexually active adolescents report using a method of contraception at some point in their lifetime - they are not typically selecting the most effective methods. Combined oral contraceptives and condoms are the most popular and most requested method of contraception by teenagers (3, 4). Unfortunately, the failure rates of both oral contraceptives and condoms among adolescents are higher compared with all typical users (5, 6). Specifically, adolescent mothers are

documented to have a high rate of repeat pregnancy and are more likely to use ineffective methods and to use effective methods inconsistently or incorrectly (6).

It is encouraging that there has been in increase in the number of adolescents who use long-acting reversible contraceptive (LARC) methods, such as the intrauterine device or contraceptive implant. With 4.5% of adolescents using such methods in 2009, compared to only 1.5% in 2007, and just 0.3% in 2002 (7). In fact, when adolescents were counseled on the full range of contraceptive options and the barrier of cost for LARC methods was removed in a large study, more than twothirds of females aged 14 – 20 years chose LARC methods (8). It is also promising that national organizations, such as the American Congress of Obstetricians and Gynecologists, have emphasized the importance of LARC method use by adolescents. Specifically, ACOG states that LARC methods are safe and appropriate for most women and adolescents, and that they provide top-tier effectiveness, high rates of satisfaction and continuation (9). Furthermore, the Contraceptive CHOICE project, a large prospective cohort study designed to promote the use of LARC methods to reduce unintended pregnancy, found that sexually active teens using the contraceptive implant or intrauterine device have significantly lower mean annual rates of pregnancy, birth, and abortion (34.0, 19.4, and 9.7 per 1000 teens) compared to sexually experienced U.S. teens (158.5, 94.0, 41.5 per 1000) (10). Data from the contraceptive CHOICE project also demonstrates that teens continued to use LARC methods longer than shorter acting methods (i.e. the oral contraceptive pill and depot medroxyprogesterone acetate injections) - two thirds of teens in the CHOICE project were still using their LARC method at 24 months, as compared with only one third of teens using a non-LARC method (11).

The sub-dermal single rod etonogestrel-only implant offers highly effective, longacting, reversible contraception (12). It consists of a single rod (4 cm in length, 2 mm in diameter) made of ethylene vinyl acetate, containing 68 mg of etonogestrel that is released subdermally over three years. Prevention of pregnancy is accomplished by several mechanisms – suppression of ovulation, thickening of

cervical mucus inhibiting sperm penetration into the uterus, and alteration of the endometrium. In the clinical trial of 301 Nexplanon (the radiopaque etonogestrel implant) users, no woman became pregnant while the implant was in situ, up to and including 14 days after implant removal. This resulted in an estimated overall Pearl Index of 0.0 (95% CI, 0.0 - 0.56) (12); which translates clinically to >99 percent effective at preventing pregnancy. They are documented to be safe for use in the adolescent population. However, the implant is currently used by less than 1% of U.S. women using contraception, and by 0.5% of those aged 15-19 years (13).

It is well documented that women using the contraceptive implant can expect changes in their menstrual bleeding patterns, and these changes account for the most commonly cited reason for method discontinuation. The bleeding pattern women experience in the first three months after insertion is predictive of future bleeding patterns throughout the duration of use (14). When analyzing 11 clinical trials, bleeding patterns were described as infrequent bleeding in 33.3% of 90-day cycles, amenorrhea in 21.4% of cycles, prolonged bleeding in 16.9% of cycles, and frequent bleeding in 6.1% of cycles (15).

There have been studies that propose management options for treating bothersome bleeding associated with the etonogestrel contraceptive implant – such options include combined oral contraceptive pills, non-steroidal anti-inflammatory agents, mefenamic acid, mifepristone, and doxycycline. Unfortunately there is limited clinical data supporting the effectiveness of these treatments (16-18). To our knowledge, there have been no studies investigating the use of oral progesterone for management of bothersome bleeding associated with the contraceptive implant. Given the success of norethindrone acetate in the management of pain and bleeding in adolescents with endometriosis (19), we chose to use norethindrone acetate as our oral progestin of choice for managing bothersome bleeding associated with the contraceptive implant.

When investigating bleeding patterns, a common challenge encountered is that of patient compliance with menstrual calendars. The burden of keeping a daily menstrual calendar may lead to reduced response rates, incomplete data, and poor data fidelity. The widespread popularity of mobile phone technology has increased the ability to connect with study participants in real time, thus decreasing the reliance on traditional pencil and paper methodology for data collection. There are several potential advantages for using short-message service text messaging (SMS) for data collection: (a) data is time stamped thus providing accurate real-time information, (b) study designers have the ability to ensure data responses conform to a set criteria, (c) automatic SMS texts provide prompts for participants to record the data of interest, (d) data transfer is instantaneous thus reducing data loss or incompleteness, and (e) data collection is more convenient and accessible for participants as they are likely to have their mobile phone devices with them and be familiar with the SMS texting function of their particular device. To our knowledge there have been no studies that use SMS text messaging to record data on daily bleeding patterns – essentially creating a real-time electronic menstrual calendar.

## **MATERIALS AND METHODS:**

We will conduct a prospective study of adolescents using the etonogestrel contraceptive implant. Participants will be recruited from the Norton Children's Gynecology practice in Louisville, Kentucky. This practice provides care to a diverse population of females, from a wide range of socioeconomic statuses, age birth to 25 years.

Inclusion criteria will include any post-menarchal female presenting to the Norton Children's Gynecology practice, who desires to use the etonogestrel contraceptive implant and has access to a mobile phone device.

All patients presenting and choosing to have an implant placed will be offered participation. The study will enroll subjects until 30 active participants are in each study arm; for a total of 60 study participants. In order to achieve the enrollment of

60 active subjects up to 100 participants will be enrolled. All enrollments will be voluntary. Participants will receive compensation for their participation. After obtaining informed consent and assent, participants will provide baseline demographic information, including: age, race/ethnicity, zip code of residence, health insurance provider, number of current and past partners, use of prior contraceptive methods, concomitant condom use, sexually transmitted infection history, age at menarche, menstrual cycle regularity, last menstrual period, weight and height. The date of etonogestrel implant insertion will be confirmed.

All patients using etonogestrel contraceptive implants will receive daily SMS texts in the evening via the Qualtrics SMS program asking them to respond with their bleeding pattern that day. If the SMS text messages are unable to connect to your personal cell phone we request an alternative cell phone number be given in order to reach you. We will record responses according to the World Health Organization definitions of bleeding: (a) bleeding day, (b) spotting day, (c) bleeding-free day [see Table I for WHO bleeding definitions]. At their initial follow-up visit 3 months after Nexplanon insertion, we will identify those who report "bothersome" bleeding patterns. For the purpose of this study, "bothersome" bleeding will be defined as prolonged and/or frequent bleeding, as characterized by World Health Organization-recommended definitions of bleeding. The definitions are listed in Table I.

| Bleeding dayAny day with vaginal discharge containing blood that required more than 1 sanitary pad or tampon per daySpotting dayAny day with vaginal discharge containing blood that required at most one sanitary pad or tampon per dayBleeding-free dayA day during which neither bleeding nor spotting was reportedBleeding-spotting episodeOne or more consecutive days during which bleeding or spotting was entered in the diary, bounded by bleeding-free daysAmenorrheaNo bleeding or spotting days throughout the 90-day reference periodInfrequent bleedingLess than three bleeding-spotting episodes in a 90-day reference period, excluding amenorrheaNormal frequencyThree to five bleeding-spotting episodes in a 90-day reference periodFrequent bleedingMore than five bleeding-spotting episodes in a 90-day reference periodProlonged bleedingAny bleeding-spotting episode (uninterrupted) lasting more than 14 days in the 90-day reference period | | |
|---|---|---|
| Bleeding-free day A day during which neither bleeding nor spotting was reported Bleeding- spotting episode Amenorrhea Infrequent bleeding Normal Frequency Frequent bleeding More than five bleeding-spotting episodes in a bleeding Prolonged A day during which neither bleeding nor spotting was reported One or more consecutive days during which bleeding or spotting was entered in the diary, bounded by bleeding or spotting days throughout the 90-day reference period Less than three bleeding-spotting episodes in a 90-day reference period, excluding amenorrhea More than five bleeding-spotting episodes in a 90-day reference period Any bleeding-spotting episode (uninterrupted) lasting more | Bleeding day | iday I I |
| Bleeding-free<br>dayA day during which neither bleeding nor spotting was reportedBleeding-<br>spotting episodeOne or more consecutive days during which bleeding or<br>spotting was entered in the diary, bounded by<br>bleeding-free daysAmenorrheaNo bleeding or spotting days throughout the<br>90-day reference periodInfrequent<br>bleedingLess than three bleeding-spotting episodes in a<br>90-day reference period, excluding amenorrheaNormal<br>frequencyThree to five bleeding-spotting episodes in a<br>90-day reference periodFrequent<br>bleedingMore than five bleeding-spotting episodes in a<br>90-day reference periodProlongedAny bleeding-spotting episode (uninterrupted) lasting more | Spotting day | Any day with vaginal discharge containing blood that required |
| A day during which neither bleeding nor spotting was reported Bleeding- spotting episode Amenorrhea No bleeding or spotting days throughout the 90-day reference period Infrequent bleeding Normal Three to five bleeding-spotting episodes in a 90-day reference period Frequent bleeding More than five bleeding-spotting episodes in a 90-day reference period More than five bleeding-spotting episodes in a 90-day reference period Any bleeding-spotting episodes (uninterrupted) lasting more | Bleeding-free | |
| spotting episodespotting was entered in the diary, bounded by bleeding-free daysAmenorrheaNo bleeding or spotting days throughout the 90-day reference periodInfrequent bleedingLess than three bleeding-spotting episodes in a 90-day reference period, excluding amenorrheaNormal frequencyThree to five bleeding-spotting episodes in a 90-day reference periodFrequent bleedingMore than five bleeding-spotting episodes in a 90-day reference periodProlongedAny bleeding-spotting episode (uninterrupted) lasting more | | A day during which neither bleeding nor spotting was reported |
| Spotting episodebleeding-free daysAmenorrheaNo bleeding or spotting days throughout the 90-day reference periodInfrequent<br>bleedingLess than three bleeding-spotting episodes in a 90-day reference period, excluding amenorrheaNormal<br>frequencyThree to five bleeding-spotting episodes in a 90-day reference periodFrequent<br>bleedingMore than five bleeding-spotting episodes in a 90-day reference periodProlongedAny bleeding-spotting episode (uninterrupted) lasting more | Bleeding- | Bleeding- One or more consecutive days during which bleeding or |
| Infrequent Less than three bleeding-spotting episodes in a 90-day reference period, excluding amenorrhea Normal Three to five bleeding-spotting episodes in a 90-day reference period Three to five bleeding-spotting episodes in a 90-day reference period Frequent Bleeding More than five bleeding-spotting episodes in a 90-day reference period Prolonged Any bleeding-spotting episode (uninterrupted) lasting more | spotting episode | |
| Description of the bleeding spotting episodes in a go-day reference period, excluding amenorrhea | Amenorrhea | |
| Normal frequency Three to five bleeding-spotting episodes in a 90-day reference period Frequent bleeding More than five bleeding-spotting episodes in a 90-day reference period Prolonged Any bleeding-spotting episode (uninterrupted) lasting more | Infrequent | |
| Three to five bleeding-spotting episodes in a 90-day reference period Frequent More than five bleeding-spotting episodes in a 90-day reference period Prolonged Any bleeding-spotting episode (uninterrupted) lasting more | bleeding | 90-day reference period, excluding amenorrhea |
| Frequent Bleeding More than five bleeding-spotting episodes in a 90-day reference period Prolonged Any bleeding-spotting episode (uninterrupted) lasting more | Normal | rmal Three to five bleeding-spotting episodes in a |
| bleeding 90-day reference period Prolonged Any bleeding-spotting episodes in a 90-day reference period | frequency | 90-day reference period |
| Prolonged Any bleeding-spotting episode (uninterrupted) lasting more | Frequent | <i>quent</i> More than five bleeding-spotting episodes in a |
| Any bleeding-spotting episode (uninterrupted) lasting more | bleeding | |
| <b>bleeding</b> than 14 days in the 90-day reference period | Prolonged | Any bleeding-spotting episode (uninterrupted) lasting more |
| | bleeding | than 14 days in the 90-day reference period |

Table I: WHO bleeding descriptions and patterns

Norethindrone acetate (aygestin) will be used to manage bothersome bleeding. Patients will be prescribed aygestin 5 mg by mouth twice daily for one month, followed by aygestin 5 mg by mouth once daily for two months. Medication will then be discontinued. Patients will be evaluated in the office three months after medication initiation, and then again six months after medication initiation. If the patient is unable to take norethindrone acetate (aygestin) due to medical contraindications or cost, they will receive medroxyprogesterone acetate (provera) 10 mg once daily as alternate oral progesterone. Figure 1 below highlights the study design.



Figure 1: Study design

During the aygestin administration, patients will again receive daily SMS texts in the evening via the Qualtrics SMS program asking them to respond with their bleeding pattern that day. We will record responses according to the World Health Organization definitions of bleeding: (a) bleeding day, (b) spotting day, (c) bleeding-free day. Patients not reporting bothersome bleeding after the initial 90 days will continue to record bleeding via SMS texts for the next 6 months to serve as the control group (normal bleeding group).

Participants will be compensated as an incentive to increase daily participation. The participant will receive a pre-paid card if they respond to >70% of text messages over each 90-day cycle and attend the scheduled office visit. Patients will receive a \$5 pre-paid card at visit one (3 months after insertion of etonorgestrel implant), \$10 pre-paid card at visit two (6 months after insertion of etonorgestrel implant), and a \$15 pre-paid card at visit three (9 months after insertion of etonogestrel implant).

At the completion of the study, 9 months after enrollment, participants will receive a SMS text message via Qualtrics with a link to a 12 question follow up survey. The post study questionnaire will assess overall satisfaction with the etonogestrel implant and evaluate participants' perceptions of text messaging as a tool to collect information. See Appendix II.

Participants who have already completed the 9 month study will receive an updated copy of the consent and assent form via mail with a request to sign the updated consent and assent forms. See Appendix III for a copy of a letter to be included with the updated consent and assent. Once the updated consent and assent are received by the investigators at Norton Children's Gynecology the post survey follow up will be sent to the participant by SMS text message via Qualtrics. Study participants who are seen in the office for their 9 month follow up visit will be re-consented in the office.

Patients diagnosed with a sexually transmitted infection during the course of the study will be removed from the study and their data will be excluded from analysis.

All completed demographic data collection forms and electronic menstrual calendars will be kept in a database, de-identified, and stored on a password-protected computer. Study size will be a convenience sample. Based on the current rate of etonogestrel implant insertions in our practice, it is anticipated that 30 participants can be recruited over a six-month period of time.

# **Data Collection and Analysis**

All patients who meet the inclusion criteria and enroll in the study will be sent a text message daily for 90 days (3 months). The daily message will prompt the participant to indicate the bleeding level for the day. This single question will have 4 options:

- 1. Bleeding Day
- 2. Spotting Day
- 3. Bleeding Free Day
- 4. Prefer not to answer today.

On day 90, descriptive tallies of the responses will be done. Using SPSS v20, an algorithm will count the number of bleeding days, spotting days, and bleeding free days and prefer not to answer (PNA) days; the data record for each participant will contain four count variables (bleeding, spotting, free, PNA). Secondly, the algorithm will identify and tally –according to WHO guidelines in Table 1 - bleeding-spotting episodes (BSE), amenorrhea (AM), infrequent bleeding (IF), normal frequency of bleeding (NF), frequent bleeding (FB), and prolonged bleeding (PB).

Participants who have at least a single episode of FB or PB will be assigned the label of "bothersome bleeding". Those without a single episode of FB or PB will be labeled "normal bleeding". Participants in the Bothersome Bleeding group will be offered aygestin to control the bothersome bleeding. Participants in the Normal Bleeding group will continue as before, with no additional medications. Following the principle of intent-to-treat, data from those in the Bothersome Bleeding group will be assigned to the aygestin group, despite that they are not taking it.

During the first month, participants in the Bothersome Bleeding group will take one 5 mg tablets of aygestin twice daily (morning and evening). After 30 days, the dose of aygestin will be halved, such that only one 5 mg tablet is taken daily. Sixty days

later, the Bothersome Bleeding group will discontinue aygestin. Ninety days later, both the normal group and the Bothersome Bleeding group will be re-evaluated.

### **Data Analysis**

A descriptive table will be used to sort participants into Normal Bleeding and Bothersome Bleeding. Non-parametric and parametric statistics will be used to compare the demographics of these two groups.

A **dose-response curve** covering six months will be plotted for the Bothersome Bleeding group to visually reveal the impact of one month of 10 mg of aygestin vs. two months of 5 mg aygestin vs. three months 0 mg of aygestin. Plotted on the curve will be the group averages of the daily bleeding value (1 for no bleeding, .5 for spotting, 0 for bleeding). A second **no-dose curve** will be added to the X-Y plot for the six months of data from the Normal Bleeding group.

Repeated Measure Multivariate Analysis of Variance (RM-ANOVA) with a Between-Subjects variable included, will be conducted (assuming sufficient data is available – e.g., low PNA rates) to compare the first 30 day average bleeding value, the 90 day bleeding average, and the 180 day bleeding average between the two groups. Planned post-hoc comparisons will evaluate changes between the control group and intervention group at the three time points.

Additional analyses may also include regression analysis to assess for predictive factors related to response to aygestin.

#### TIMELINE:

October 2014 IRB Submission

November 2014 Anticipated IRB Approval

November 2014 –

July 2015

**Data Collection** 

August – September 2015 Data Analysis

October 2015 Submission of preliminary data to the North

American Society for Pediatric and Adolescent Gynecology (NASPAG) Annual Clinical and

Research Meeting Board

April 2016 Present at the North American Society for

Pediatric and Adolescent Gynecology (NASPAG)

Annual Clinical and Research Meeting

May 2016 Final manuscript composition and submission

for publication

### **APPENDICES:**

Appendix I: Demographic Data Collection Form

## **INFORMED CONSENT / ASSENT:**

See the attached University of Louisville Biomedical Informed Consent and Assent Forms.

#### **REFERENCES:**

- 1. Finer LB, Aolna MR. Unintended pregnancy in the United States: incidence and disparities, 2006. Contraception 2011; 84:478-85.
- 2. The Alan Guttmacher Institute. U.S. Teenage Pregnancy Statistics. National and State Trends and Trends by Race and Ethnicity, 2006, The Alan Guttmacher Institute, New York, 2009.
- 3. The Alan Guttmacher Institute. U.S. Teenage Pregnancy Statistics. National and State Trends and Trends by Race and Ethnicity, 2006, The Alan Guttmacher Institute, New York, 2009.
- 4. Abma JC, Martinez GM, Copen CE. Teenagers in the United States: sexual activity, contraceptive use, and child bearing. National Survey of Family Growth 2006-2008. National Center for Health Statistics. Vital Health Stat 23 2012;(30):1-47.
- 5. Fu H, Darroch JE, Haas T, Ranjit N. Contraceptive failure rates: new estimates from the 1995 National Survey of Family Growth, Fam Plann Perspect 31: 58, 1999.
- 6. Speroff L, Darney PD. A Clinical Guide for Contraception, 5<sup>th</sup> ed. 11: 360, 2011.
- 7. Finer LB, Jerman J, Kavanaugh MD. Changes in the use of long-acting contraceptive methods in the United States, 2007-2009. Fertil Steril 2012; 98(4):893-97.
- 8. Mestad R, Secura G, Allsworth JE, Madden T, Zhao Q, Peipert JF. Acceptance of long-acting reversible contraceptive methods by adolescent participants in the Contraceptive CHOICE Project. Contraception 2011; 84:493-8.
- 9. "Adolescents and Long-Acting Reversible Contraception: Implants and Intrauterine Devices." American College of Obstetricians and Gynecologists Committee Opinion #539. October 2012.
- 10. Secura GM, Maden T, McNichols C, et al. Provision of no-cost, long-acting contraception and teenage pregnancy. N Engl J Med 2014; 371:1316-23.
- 11. O'Neil-Callahan M, Peipert JF, Zhao Q, et al. Twenty-four month continuation of reversible contraception. Obstet Gynecol 2013; 122:1083-91.
- 12. Mommers E, Blum G-F, Gent TG, et al. Nexplanon, a radiopaque etonogestrel implant in combination with a next-generation applicator: 3 year results of a noncomparative multicenter trial. Am J Obstet Gynecol 2012; 207:388.e1-6.
- 13. Mosher WD, Jones J. Use of contraception in the United States: 1982 2008. Vital Health Stat 23 2010; (29): 1-44.
- 14. Monsour, D, Korver T, Marintcheva-Petrova M, Fraser IS. The effects of Implanon on menstrual bleeding patterns. Eur J Contracept Reprod Health Care 2008; 13(suppl 1): 12-28.
- 15. Darney P, Patel A, Rosen K, Shapiro LS, Kaunitz AM. Safety and efficacy of a single-rod etonogestrel implant (Implanon): results from 11 international clinical trials. Fertil Steril 2009;91:1646-53.
- 16. Mansour D, Bahamondes L, Critchley H, Darney P, Fraser IS. The management of unacceptable bleeding patterns in etonogestrel-releasing contraceptive

- implant uses. Contraception 2011;83:202-10.
- 17. Phaliwong P, Taneepanichskul S. The effect of mefanamic acid on controlling irregular uterine bleeding second to Implanon Use. J Med Assoc Thai 204;87(suppl 3):S64-8.
- 18. Weisberg E, Hickey M, Palmer D, O'Connor V, Salamonsen LA, Findlay JK, et al. A randomized controlled trial of treatment options for troublesome uterine bleeding in Implanon users. Hum Reprod 2009;24:1852-61.
- 19. Kaser DJ, Missmer SA, Berry KF et al. Use of norethindrone acetate alone for postoperative suppression of endometriosis symptoms. J Pediatr Adolesc Gynecol 2012; 25:105-108.

# APPENDIX I:

## **DEMOGRAPHIC DATA COLLECTION FORM:**

| What is your age? Years old | Are you currently using condoms? Most / All of the time Some of the time |
|---|---|
| | None of the time |
| Are you Hispanic or Latino? | |
| Yes, Hispanic or Latino | |
| No, not Hispanic or Latino | Have you ever had a sexually transmitted infection? |
| | Chlamydia |
| How would you describe yourself? | Gonorrhea |
| Choose one or more from the following | Trichomonas |
| ethnic/racial groups: | Herpes |
| American Indian or Alaskan Native | HIV / AIDS |
| Asian | Hepatitis B |
| Black or African American | Hepatitis C |
| Native Hawaiian or Pacific Islander White | Syphilis |
| What is your zip code? | How old were you when you started having periods? |
| | Years old |
| Health insurance provider | Are you currently having a monthly |
| Private insurance | menstrual cycle? |
| Medicaid (i.e. passport) | Yes |
| No insurance | No |
| Sexual partners | What was the first day of your last |
| In the past month In your lifetime | menstrual period? |
| Use of prior contraceptive methods | What is your weight? |
| Pills | Pounds |
| Patch | |
| Ring | |
| Depo-Provera | What is your height? |
| Intrauterine device | Inches |
| Condoms | _ |
| Spermicide | |
| Sponge | When was your implant put in? |
| Diaphragm | Date |
| Withdrawal | _ |

# Appendix II:

| 1 | How do you feel about using text messages as a way of telling the researchers about your period or break-through bleeding? | Very happy | Нарру | Neutral | Un-happy | Very Un-<br>happy |
|---|---|---|---|---|---|---|
| 2 | Did you answer the text messages every day? | All of the time | Most of the time | Some of the time | Hardly<br>ever | Never [1] |
| 3 | When you were not able to answer the text message, what were the reasons for not doing so? Choose all that apply | Busy doing<br>some-thing<br>else | Forgot<br>about to<br>answer | Lost<br>access to<br>my phone | Ran out<br>of<br>minutes/<br>texts | Other |
| 4 | Did you ever feel annoyed or unhappy about receiving texts from the researchers? | No, never | Rarely | Some-<br>times | About<br>once a<br>week | Every day |
| 5 | Would you be more or less likely to enroll in a future study if that study also used text messages to collect your information? | Much less<br>likely to<br>enroll | Less<br>likely to<br>enroll | Makes No<br>differ-<br>ence | More<br>likely to<br>enroll | Much more<br>likely to<br>enroll |
| 6 | Text messages were sent at 6pm every evening. How did you feel about the timing of the texts? | | Better<br>earlier in<br>the day | The<br>timing<br>was fine | Better<br>later in<br>the day | |
| 7 | For this type of research, another way of collecting data is to have you write your information into a paper-based diary each day. Which method of data collection would you prefer? | Strongly<br>prefer<br>paper-<br>based diary | Prefer<br>paper<br>based<br>diary | Either<br>would be<br>fine | Prefer<br>text-<br>based | Strongly<br>prefer text-<br>based |
| 8 | Throughout the study period (up to 270 days), how often did you change your cell phone plan (for example, get a new phone number, change your plan to get more or fewer messages, etc.)? | Never | 1 time | 2 times | 3 times | More than 3 times |
| 9 | Did the text message format make it easier or harder for you to give your answer truthfully? | Much<br>Easier | Easier | No differ-<br>ence | Harder | Much<br>Harder |
| 10 | How likely do you think your friends would be willing to enroll in a study that uses text messaging for collecting data? | Very likely | Likely | Neither<br>likely nor<br>unlikely | Unlikely | Very<br>unlikely |
| 11 | Do you plan to keep your<br>Nexplanon for the next 9 months or<br>longer? | Already<br>removed it | No | Un-<br>decided | Yes | |
| 12 | Would you recommend Nexplanon to a friend? | Definitely<br>no | Maybe<br>no | Undecide<br>d | Maybe<br>yes | Definitely<br>yes |

# Appendix II:

| 1 | How do you feel about using text messages as a way of telling the researchers about your period or break-through bleeding? | Very happy | Нарру | Neutral | Un-happy | Very Un-<br>happy |
|---|---|---|---|---|---|---|
| 2 | Did you answer the text messages every day? | All of the time | Most of the time | Some of the time | Hardly<br>ever | Never |
| 3 | When you were not able to answer the text message, what were the reasons for not doing so? Choose all that apply | Busy doing<br>some-thing<br>else | Forgot<br>about to<br>answer | Lost<br>access to<br>my phone | Ran out<br>of<br>minutes/<br>texts | Other |
| 4 | Did you ever feel annoyed or unhappy about receiving texts from the researchers? | No, never | Rarely | Some-<br>times | About<br>once a<br>week | Every day |
| 5 | Would you be more or less likely to enroll in a future study if that study also used text messages to collect your information? | Much less<br>likely to<br>enroll | Less<br>likely to<br>enroll | Makes No<br>differ-<br>ence | More<br>likely to<br>enroll | Much more<br>likely to<br>enroll |
| 6 | Text messages were sent at 6pm every evening. How did you feel about the timing of the texts? | | Better<br>earlier in<br>the day | The<br>timing<br>was fine | Better<br>later in<br>the day | |
| 7 | For this type of research, another way of collecting data is to have you write your information into a paper-based diary each day. Which method of data collection would you prefer? | Strongly<br>prefer<br>paper-<br>based diary | Prefer<br>paper<br>based<br>diary | Either<br>would be<br>fine | Prefer<br>text-<br>based | Strongly<br>prefer text-<br>based |
| 8 | Throughout the study period (up to 270 days), how often did you change your cell phone plan (for example, get a new phone number, change your plan to get more or fewer messages, etc.)? | Never | 1 time | 2 times | 3 times | More than 3 times |
| 9 | Did the text message format make it easier or harder for you to give your answer truthfully? | Much<br>Easier | Easier | No differ-<br>ence | Harder | Much<br>Harder |
| 10 | How likely do you think your friends would be willing to enroll in a study that uses text messaging for collecting data? | Very likely | Likely | Neither<br>likely nor<br>unlikely | Unlikely | Very<br>unlikely |
| 11 | Do you plan to keep your<br>Nexplanon for the next 9 months or<br>longer? | Already<br>removed it | No | Un-<br>decided | Yes | |
| 12 | Would you recommend Nexplanon to a friend? | Definitely<br>no | Maybe<br>no | Undecide<br>d | Maybe<br>yes | Definitely<br>yes |

#### Appendix III:

Norton Children's Gynecology 3991 Dutchmans Lane, Suite 303 Louisville, KY 40207

Dear Study Participant,

You had participated in an etonogestrel contraceptive implant (Nexplanon) study for 9 months. We have created a 12-question follow up survey to evaluate your satisfaction with the Nexplanon and your perception of text messaging as a tool to collect information. We would like to send you a text message with a link to the post study survey.

Enclosed you will find an updated copy of the Consent and Assent forms. You had completed these Consent and Assent forms in the office 9 months ago. These updated documents however now include information about the 12-question follow up survey. The Consent is updated on page 2, paragraph 5 and the Assent is updated in paragraph 4. Prior to sending you a text message link to the post study survey both the Consent and Assent forms will need to be signed and mailed back to our office.

We would appreciate if you could please read the documents and then have the participant's guardian sign the Consent form on page 8 and the study participant sign the Assent form on Page 2. These documents can then be placed in the enclosed return envelope and mailed to our office.

Thank you for your participation in the study as we value your input. Should you have any questions about the survey or enclosed documents please call our office to speak with study personnel at (502) 559-1750.

Thank you,

Rachael Polis, DO